CLINICAL TRIAL: NCT06758921
Title: Prospective, Multicenter, Single-Arm Observational Study to Confirm the Safety and Clinical Performance of the Oscar Peripheral Multifunctional Catheter for the Dilatation of Lesions in the Femoral, Popliteal and Infrapopliteal Arteries
Brief Title: Prospective, Multicenter, Single-Arm Observational Study to Confirm the Safety and Clinical Performance of the Oscar Peripheral Multifunctional Catheter for the Dilatation of Lesions in the Femoral, Popliteal and Infrapopliteal Arteries (BIO-OSCAR First)
Status: Recruiting | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C2401
Record Dates: First submitted 2024-10-31; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Arterial Disease; Peripheral Arterial Disease(PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Oscar Peripheral Multifunctional Catheter — Oscar Peripheral Multifunctional Catheter encompasses three components: (i) Oscar Support Catheter with integrated Lock Grip, (ii) Oscar Dilator and (iii) Oscar PTA Balloon.
  Single Oscar PTA Balloon is also available separately and can only be used together with the pre-supplied Oscar Support Catheter as indicated in the compatibility chart in the Instructions for Use (IFU).

SUMMARY:
The purpose of this study is to evaluate the standard of care practices, procedural outcomes, and in-hospital complications for endovascular peripheral interventions of femoral, popliteal and infrapopliteal lesions.

DETAILED DESCRIPTION:
This is a prospective, multicenter, all-comers observational study. Primary endpoint was procedural success (defined as a combination of successful primary target lesion crossing, residual stenosis of ≤30% following vessel preparation and before definite treatment) and absence of procedural complications (defined as target vessel perforation or rupture, acute occlusion, and distal embolization).

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥18 years old
2. Subject has provided written informed consent
3. Subject has Rutherford classification 2 to 6
4. Reference vessel diameter ≥2 and ≤7 mm
5. Target lesion(s) has stenosis >70% by visual assessment
6. Multiple consecutive single lesions with a healthy segment(s) of ≤ 3cm in-between will be considered one lesion.

   Above the knee (ATK) group:
7. Target lesions located in the superficial femoral artery or popliteal arteries (above the tibial plateau)
8. At least one below-knee artery patent to the ankle
9. Successful treatment of inflow iliac stenosis to the target lesion. Inflow lesion stenosis can be treated during the same procedure as per local standard of care. The inflow lesion(s) must be treated first, prior to consideration of treatment of the target lesion. Subject can be enrolled if the inflow lesion(s) are treated and result in ≤30% residual stenosis and no evidence of embolization or significant complications.

   Below the knee (BTK) group:
10. Target lesions involve arteries below the tibial plateau
11. Successful treatment of inflow vessel (from ipsilateral iliac to the target lesion) resulting in ≤30% residual stenosis with no evidence of embolization or significant complications

Exclusion Criteria:

1. Subject has a single target lesion that involves both ATK and BTK segments.
2. Subject not suitable for receiving endovascular procedures of lower limb arteries.
3. Prior planned major amputation in the target limb (i.e., above the ankle).
4. Subject with previous bypass surgery of target vessel.
5. History of any open surgical procedure within the past 30 days.
6. Planned vascular surgery procedure within the next 30 days after the ATK and/or BTK procedure on the target limb.

   Note: The inflow vessels can be treated on the day of the procedure.
7. Subject has Oscar IFU listed contraindication (such as uncorrected bleeding disorders, sepsis).
8. Subject under dialysis.
9. Subject currently enrolled in another investigational device, biologic, or drug trial in which the primary endpoint has not yet been reached.
10. Subject lacking capacity to provide informed consent.
11. Subject under judicial protection, tutorship, or curatorship (for France only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 200 patients will be enrolled, with approximately 100 subjects in ATK group, and 100 subjects in BTK group.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Oscar Procedural success rate | Index procedure
  combination of Oscar technical success and absence of serious procedural complications

SECONDARY OUTCOMES:
Rate of (Serious) Adverse Device Effects (S)ADE | discharge (30 days)
  (Serious) Adverse Device Effects
Rate of distal embolization | Index procedure
  Distal embolization
Rate of target vessel rupture | Index procedure
  Target vessel rupture
Rate of target vessel perforation | Index procedure
  Target vessel perforation
Rate of target vessel acute occlusion | Index procedure
  Target vessel acute occlusion
Rate of Oscar PTA balloon related flow-limiting dissections | Index procedure
  flow-limiting dissections defined as NHLBI grade ≥D
Rate of peri-operative death (all-cause of death until discharge) | discharge (30 days)
  peri-operative death defined as all-cause of death until discharge
Rate of unplanned major amputation | discharge (30 days)
  unplanned major amputation
Oscar crossing success | Index procedure
  angiographic confirmation of successful placement of a guidewire into the distal true lumen with Oscar support catheter used together with the dilator and/ or Oscar PTA balloon, and without any additional crossing/re-entry device.
Post-Oscar residual stenosis | Index procedure
  Post-Oscar residual stenosis (%)
Final treatment residual stenosis (%) on the completion angiogram | Index procedure
  Final residual stenosis (%) on the completion angiogram

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, Principal Investigator — AZ Saint Blasius
Locations (16):
- LKH Univ. -Klinikum Graz, Ambulanz für Angiologie, Graz, Austria
- Belgium (5):
  - Onze Lieve Vrouwziekenhuis, Aalst
  - AZ Saint Blasius, Dendermonde
  - ZOL Ziekenhuis Oost Limburg, Genk
  - University Hospital Ghent, Ghent
  - vzw AZ Groeninge, Kortrijk
- Hopital Saint Joseph, Paris, France
- Germany (3):
  - Karolinen-Hospital Arnsberg, Arnsberg
  - Sankt Gertrauden-Krankenhaus, Berlin
  - Universitätsklinikum Tübingen, Tübingen
- Semmelweis University, Budapest, Hungary
- Italy (3):
  - Policlinico Abano Terme, Abano Terme
  - Azienda Usl Toscana sud est, Arezzo
  - ospedaliero-universitaria Senese, Siena
- Hospital Universitario de Guadalajara, Guadalajara, Spain
- Ospedale Regionale civico EOC di Lugano, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided